CLINICAL TRIAL: NCT02797314
Title: Comparison of Bone Quality in Type 2 Diabetic Patients With a Non-diabetic Control Population
Acronym: DIABONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL16_0092; 2016-A01228-43 (Other: ANSM)
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Bone quality; Bone biopsies; Vertebral fractures; Osteodensitometry; Trabecular Bone Score
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetic population (Other): Bone biopsies
  Interventions: Other: Bone biopsies
- Non-diabetic control population (Other): Bone biopsies
  Interventions: Other: Bone biopsies

INTERVENTIONS:
Other: Bone biopsies — Bone biopsies

SUMMARY:
Patients with type 2 diabetes have many complications in different organs. These complications are extremely frequent and severe: cardiovascular and renal disease, visual impairment, and, more recently, complications affecting bone such as fractures. Conventional methods for the evaluation of fracture risk are based on the Bone Mineral Density (BMD) or FRAX (algorithm for the prediction of osteoporotic fracture risk) are not sufficient in the context of diabetes. Several metaanalyses have shown that, paradoxically, a higher BMD in patients with type 2 diabetes compared to patients not suffering from this disease, independently of body mass index (BMI). The paradoxal increase in fracture risk, despite a high BMD has led to the hypothesis that diabetes induces a modification of the quality and not the quantity of bone. However, there is a lack of data as to bone quality in patients with type 2 diabetes as studies of bone biopsies from patients with type 2 diabetes are extremely rare.

The objective of the study is to compare bone quality in patients with type 2 diabetes to that in patients who do not suffer from type 2 diabetes: evaluation of vertebral fractures by osteodensitometry, measurement of Trabecular Bone Score (TBS), and analysis of bone quality in biopsies (advanced glycation end products (AGE), contents of bone matrix and analysis of mineralization).

The results will then be correlated with blood/urinary markers with the objective to determine one/several non-invasive biomarkers for bone status in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged greater than 40 years
* Patients requiring surgery of the lower limb
* With a bone mineral density considered normal (T-score ≥ -2)
* Stage 1, 2, or 3 glomerular filtration rate (> 30 mL/min)
* For diabetic patients the diagnosis will have previously established by an endocrinologist

Exclusion Criteria:

* Subjects treated with drugs known to interfere with bone metabolism, including steroids, anticonvulsants, diuretics, and bisphosphonates
* Patients with severe renal disease (< 30 ml/mn); previous history of caner except skin cancer; myocardial infarction; uncontrolled hypertension; untreated hyperthyroidism; hyperthyroidism; malabsorption; bone metabolism diseases; rheumatoid arthritis or collagen diseases
* Pregnant or lactating woman
* Contraindication to taking tetracycline hydrochloride:

  * Known hypersensitivity to antibiotics of the tetracycline family or any of the excipients in the medicine
  * Severe chronic renal failure
  * Chronic liver failure
  * Systemic lupus erythematosus
  * Concomitant prescription of retinoid or vitamin A (risk intracranial hypertension)
* Psychiatric pathology seriously hampering understanding
* Difficulty understanding oral French
* Not a beneficiary of a social security scheme

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 1 month after patient inclusion
  Bone mineral density (BMD) measured by Dual-energy X-ray absorptiometry (DXA)
Vertebral fractures | 1 month after patient inclusion
  Presence of vertebral fractures evaluated by Vertebral Fracture Assessment (VFA)
Trabecular Bone Score | 1 month after patient inclusion
  Trabecular bone score (TBS) is a analytical tool that performs novel grey-level texture measurements on lumbar spine dual X-ray absorptiometry (DXA) images, and thereby captures information relating to trabecular microarchitecture

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Hospices Civisl de Lyon, Lyon, France